CLINICAL TRIAL: NCT05560490
Title: Safety and Performance of FibroFix™ Cartilage P Implant and Drill Set for Articular Cartilage Repair Within the Knee Joint
Brief Title: FibroFix Cartilage P Knee Implant Study
Acronym: FFLEX
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Safety issues
Sponsor: Orthox Limited (Industry)
Collaborators: Avania B.V. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORTH CIP A001
Record Dates: First submitted 2022-09-18; First posted 2022-09-29 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Osteoarthritis, Knee
Keywords: knee; cartilage repair; articular cartilage lesion; Cartilage implant
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: multicentre, prospective, non-randomised, open-label, first-in-human
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FibroFix Cartilage P Implant + Drill set (Experimental): Participants that have been implanted with FibroFix Cartilage P Implant using the FibroFix Drill Set
  Interventions: Device: FibroFix Cartilage P Knee Implantation

INTERVENTIONS:
Device: FibroFix Cartilage P Knee Implantation — The FibroFix Cartilage P instrument set (Drill set) is used for the preparation of an implant site and placement of the FibroFix Cartilage P Implant to resurface an articular cartilage lesion in the anterior and central regions of the femoral condyles of the knee.

SUMMARY:
This is a multi-center first-in-human prospective clinical investigation to evaluate the safety and performance of the FibroFix™ Cartilage P Implant and Drill Set. The Implant is a medical device designed by Orthox Ltd. to repair a damaged area of cartilage within the knee joint.

The aim is to 75 participants over two Stages:

In STAGE I, up to a total of 6 subjects will be recruited and safety assessed after 6 months of follow-up.

In Stage II an additional 69 subjects. The subjects will be followed up for 2 years with MRI imaging, then a further 8 years with patient outcome questionnaires.

DETAILED DESCRIPTION:
This is a multi-center, prospective, non-randomized, open-label clinical investigation. Safety oversight throughout will be provided by an independent data monitoring committee (DMC). The clinical investigation will be split into two stages.

Stage I of the clinical investigation will enroll a small cohort of subjects, up to a total of 6 (accounting for a 17% dropout rate) having been implanted with the FibroFix Cartilage P, to provide a minimum of 5 evaluable subjects. The initial safety of the FibroFix Cartilage P implant and the FibroFix Cartilage P Drill Set will be evaluated in these subjects across a maximum of 2 sites. Recruitment into the clinical investigation will then be paused.

Following the implantation of FibroFix Cartilage P in the initial cohort of subjects, the DMC will monitor all emerging safety issues against the stopping rules of the clinical investigation. Any treatment-emergent Serious Adverse Events (SAE) or other safety concerns during Stage I of the clinical investigation will immediately be referred, on a case-by-case basis, to the DMC for review against the stopping rules.

A formal review of safety against the stopping rules will be undertaken by the DMC at two-time points:

1. when all of the initial cohort of subjects complete 3 months post-surgery follow-up;
2. when all of the initial cohort of subjects complete 6 months post-surgery follow-up.

Each DMC review will be triggered by the last subject within the safety cohort completing the relevant 3-month and 6- month post-surgery follow-up activities, respectively.

The re-opening of recruitment will only be triggered by authorization from the DMC to proceed.

Stage II of the clinical investigation will evaluate the performance and safety of FibroFix Cartilage P and the FibroFix Cartilage P Drill Set in a wider group of subjects, a further 69 recruited from all participating clinical centers to provide 60 evaluable out of 75 recruited subjects who have been implanted with the FibroFix Cartilage P, allowing for 20% drop out rate.

Stage I (safety cohort) subjects will be analyzed with the Stage II subjects as an overall cohort unless amendments to the treatment protocol and/or medical device are required following the evaluation of the safety cohort.

Primary outcomes will be reported in an interim report following completion of the 1-year post-surgery follow-up. All subjects will be follow-up for a total of 2 years post-surgery after which a final clinical study report will be written.

All participants in this clinical investigation will receive a single appropriately sized FibroFix Cartilage P implant, surgically implanted using the corresponding FibroFix Cartilage P Drill Set.

If it is not possible to implant FibroFix Cartilage P during surgery because the lesion is too large or, if once debrided the area is too large for study implant, the standard of care will be implemented at the discretion of the surgeon, and any adverse events related to use of the FibroFix cartilage P Drill Set will be followed.

The objective of Stage I, the initial safety cohort, will be to demonstrate the safety of FibroFix Cartilage P implant in a small number of subjects at 3- and 6-month post-surgery follow-up, and FibroFix Cartilage P Drill Set intraoperatively.

The objective of Stage II, Full cohort, will be to demonstrate the performance and safety of FibroFix Cartilage P implant at 1-year post-surgery follow-up, and FibroFix Cartilage P Drill Set intraoperatively. Performance of FibroFix Cartilage P will be determined by change in the Knee Injury and Osteoarthritis Outcome Score (KOOS) Pain and Function (Sport/Rec) scores from baseline at 1-year post-surgery follow-up.

The null hypothesis being tested is the mean improvement in KOOS pain score at 1-year post-surgery from baseline is less than or equal to 8 points versus the alternative hypothesis that the mean improvement is greater than 8 points.

Subject participation will last 2 years and will require several visits to the doctor's office. Screening:

Subjects who are potential candidates for the clinical investigation will be identified by clinical research team members at the clinical centers involved. During the Screening phase, the following assessments will be performed:

* Collection of informed consent;
* Eligibility checked with subject against inclusions and exclusion criteria; • Collection of demographic and medical history data;
* Magnetic Resonance imaging (MRI).

Pre-operative Assessment:

If the subject has consented to participate and meets the inclusion criteria but none of the exclusion criteria, the following baseline assessments will be conducted. The subject's following medical history and medication history will be reviewed as part of this baseline assessment: demographics, patient history, and physical (review of systems, allergies, vital signs, physical examination, MRI assessment available to provide diagnosis, and urine pregnancy test for female subjects), concomitant medications, and MRI will be reviewed and baseline questionnaires (KOOS, Lysholm Knee Score and Tegner Activity Scale, Visual Analogue Scale (VAS) Pain, EuroQol 5-Dimension 5-Level (EQ-5D-5L), and Kellgren and Lawrence system) will be completed.

Post-operative Assessment:

For the study, subjects have to visit the hospital 6 times over 2 years (at 2w, 6w, 3m, 6m, 1y, and 2y). During all the follow-up visits, concomitant medications and safety events will be reviewed and subjects have to complete the VAS Pain, Lysholm, and Tegner activity questionnaires. In addition, during all visits except the 2w visit, subjects have to complete the KOOS questionnaire. During the 6m, 1y, and 2y visits, patients also have to complete the EQ-5D. An MRI will be conducted at 3m, 6m, 1y, and 2y.

Participants will then be followed up for a further 8 years for Device related adverse events and the same patient outcome questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is able to provide written informed consent;
2. Age ≥18 years at time of enrolment;
3. Able to comply with the protocol-defined pre-operative procedures, the post-operative clinical and imaging evaluations and the recommended rehabilitation regimen as determined by the Investigator;
4. Has a joint surface lesion, ICRS Grade 3 or above, on femoral condyles;
5. Female subjects of child-bearing potential: a negative urine pregnancy test at time of enrolment.
6. Patient has been diagnosed by MRI or other imaging technique to confirm presence of cartilage lesion and the lesion remains symptomatic. Only patients for whom the decision to perform surgery has already been made will be invited to participate. Asymptomatic lesions will NOT be included;

   Intra-Operative Inclusion criterion:
7. Lesion area of less than of 26.6 mm height and less than 20.0 mm width in the index knee after debridement.

Exclusion Criteria:

1. Age >65 years or <18 years at time of enrolment;
2. Body Mass Index (BMI) > 35;
3. Lesion area of more than 26.6 mm length and more than 20.0 mm width in the index knee after debridement;
4. Patient has multiple lesions to be treated;
5. Articular cartilage lesions in the tibia or patella, ICRS grades 3 and above;
6. KOOS Pain Subscale score at baseline that is < 20 or > 65. (Scale range: Maximum pain = 0, pain free = 100);
7. Patient has previously received the FibroFix™ Cartilage P implant;
8. Patient suffers from any medical condition that would hinder cartilage repair, such as additional unresolved comorbidities related to the index knee;

   1. Clinically significant untreated ligament instability of the same knee,
   2. Patient is post op from surgery on the same knee within 6 months which stipulates on-going rehabilitation,
   3. Untreated, symptomatic, unstable meniscal lesions on patients with residual meniscus volume of <50% in the same compartment,
   4. Joint malalignment that in the opinion of the treating surgeon, requires osteotomy to correct,
   5. Any previous surgical cartilage treatment in the index knee within the previous 6 months,
   6. Evidence of osteonecrosis of the involved knee.
9. A known allergy to:

   1. General and/or regional anaesthetic,
   2. Silk or silk containing products, or
   3. Glycerol or products containing glycerol.
10. Demonstrating an active local or systemic infection;
11. Any condition, which in the judgment of the Investigator would preclude adequate evaluation of the FibroFix™ Cartilage P implant and clinical outcome;
12. A history of confirmed anaphylactoid reaction;
13. Has received local administration of any type of corticosteroid or systemic administration of antineoplastic, immunostimulating, or immunosuppressive agents within 180 days prior to the scheduled surgery;
14. Medical history that includes a confirmed diagnosis of rheumatoid or inflammatory arthritis, or relapsing polychondritis;
15. If female and of child-bearing potential: evidence of a positive pregnancy test or a stated intention to become pregnant in the next 6 months at time of enrolment;
16. Currently participating in another device or drug clinical investigation or has done so in the previous 3 months which would impact the results of the surgery in the opinion of the surgeon or be a barrier to participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
Change in Knee injury and Osteoarthritis Outcome score (KOOS) - year 1(Pain and Sport/Rec only) | baseline (pre-surgery) to 1 year after surgery
  The knee injury and Osteoarthritis Outcome Score is a patient-assessed outcome score. Questions use a 5-point Likert scale response. KOOS is scored into 5 subscales; Pain, other Symptoms, Activities of Daily Living (ADL) Sport and Recreation Function (Sport/Rec), and knee-related quality of life (QoL). Each subscale ranges from 0 indicating extreme symptoms to 100 indicating no symptoms. Subscale scores will be aggregated and averaged as a primary outcome.
  Change from baseline of 8 points in KOOS Pain scores and Function (Sport/Rec) scores at 1-year post-surgery.
Safety endpoint - year 1 | up to year 1 after surgery
  Incidence of device related Adverse Events

SECONDARY OUTCOMES:
Change in KOOS -week 6 | baseline (pre-surgery) to week 6 after surgery
  Knee injury and Osteoarthritis Outcome Score is a patient assessed outcome score. Questions use a 5 point Likert scale response. KOOS is scored into 5 subscales; Pain, other Symptoms, Activities of Daily Living (ADL) Sport and Recreation Function (Sport/Rec) and knee-related quality of life (QoL). Each subscale ranges from 0 indicating extreme symptoms to 100 indicating no symptoms. Subscale scores will be aggregated and averaged as a primary outcome. The primary analysis repeated measures mixed model will be used to obtain estimates for additional time points as secondary objectives. Changes from baseline of mean subscale scores plotted over time to visualise change.
Change in KOOS -month 3 | baseline (pre-surgery) to month 3 after surgery
  Knee injury and Osteoarthritis Outcome Score is a patient assessed outcome score. Questions use a 5 point Likert scale response. KOOS is scored into 5 subscales; Pain, other Symptoms, Activities of Daily Living (ADL) Sport and Recreation Function (Sport/Rec) and knee-related quality of life (QoL). Each subscale ranges from 0 indicating extreme symptoms to 100 indicating no symptoms. Subscale scores will be aggregated and averaged as a primary outcome. The primary analysis repeated measures mixed model will be used to obtain estimates for additional time points as secondary objectives. Changes from baseline of mean subscale scores plotted over time to visualise change.
Change in KOOS -month 6 | baseline (pre-surgery) to month 6 after surgery
  Knee injury and Osteoarthritis Outcome Score is a patient assessed outcome score. Questions use a 5 point Likert scale response. KOOS is scored into 5 subscales; Pain, other Symptoms, Activities of Daily Living (ADL) Sport and Recreation Function (Sport/Rec) and knee-related quality of life (QoL). Each subscale ranges from 0 indicating extreme symptoms to 100 indicating no symptoms. Subscale scores will be aggregated and averaged as a primary outcome. The primary analysis repeated measures mixed model will be used to obtain estimates for additional time points as secondary objectives. Changes from baseline of mean subscale scores plotted over time to visualise change.
Change in KOOS -year 1 | baseline (pre-surgery) to year 1 after surgery
  Knee injury and Osteoarthritis Outcome Score is a patient assessed outcome score. Questions use a 5 point Likert scale response. KOOS is scored into 5 subscales; Pain, other Symptoms, Activities of Daily Living (ADL) Sport and Recreation Function (Sport/Rec) and knee-related quality of life (QoL). Each subscale ranges from 0 indicating extreme symptoms to 100 indicating no symptoms. Subscale scores will be aggregated and averaged as a primary outcome. The primary analysis repeated measures mixed model will be used to obtain estimates for additional time points as secondary objectives. Changes from baseline of mean subscale scores plotted over time to visualise change.
Change in KOOS -year 2 | baseline (pre-surgery) to year 2 after surgery
  Knee injury and Osteoarthritis Outcome Score is a patient assessed outcome score. Questions use a 5 point Likert scale response. KOOS is scored into 5 subscales; Pain, other Symptoms, Activities of Daily Living (ADL) Sport and Recreation Function (Sport/Rec) and knee-related quality of life (QoL). Each subscale ranges from 0 indicating extreme symptoms to 100 indicating no symptoms. Subscale scores will be aggregated and averaged as a primary outcome. The primary analysis repeated measures mixed model will be used to obtain estimates for additional time points as secondary objectives. Changes from baseline of mean subscale scores plotted over time to visualise change.
Change in KOOS -year 3 | baseline (pre-surgery) to year 3 after surgery
  Knee injury and Osteoarthritis Outcome Score is a patient assessed outcome score. Questions use a 5 point Likert scale response. KOOS is scored into 5 subscales; Pain, other Symptoms, Activities of Daily Living (ADL) Sport and Recreation Function (Sport/Rec) and knee-related quality of life (QoL). Each subscale ranges from 0 indicating extreme symptoms to 100 indicating no symptoms. Subscale scores will be aggregated and averaged as a primary outcome. The primary analysis repeated measures mixed model will be used to obtain estimates for additional time points as secondary objectives. Changes from baseline of mean subscale scores plotted over time to visualise change.
Change in KOOS -year 4 | baseline (pre-surgery) to year 4 after surgery
  Knee injury and Osteoarthritis Outcome Score is a patient assessed outcome score. Questions use a 5 point Likert scale response. KOOS is scored into 5 subscales; Pain, other Symptoms, Activities of Daily Living (ADL) Sport and Recreation Function (Sport/Rec) and knee-related quality of life (QoL). Each subscale ranges from 0 indicating extreme symptoms to 100 indicating no symptoms. Subscale scores will be aggregated and averaged as a primary outcome. The primary analysis repeated measures mixed model will be used to obtain estimates for additional time points as secondary objectives. Changes from baseline of mean subscale scores plotted over time to visualise change.
Change in KOOS -year 5 | baseline (pre-surgery) to year 5 after surgery
  Knee injury and Osteoarthritis Outcome Score is a patient assessed outcome score. Questions use a 5 point Likert scale response. KOOS is scored into 5 subscales; Pain, other Symptoms, Activities of Daily Living (ADL) Sport and Recreation Function (Sport/Rec) and knee-related quality of life (QoL). Each subscale ranges from 0 indicating extreme symptoms to 100 indicating no symptoms. Subscale scores will be aggregated and averaged as a primary outcome. The primary analysis repeated measures mixed model will be used to obtain estimates for additional time points as secondary objectives. Changes from baseline of mean subscale scores plotted over time to visualise change.
Change in KOOS -year 6 | baseline (pre-surgery) to year 6 after surgery
  Knee injury and Osteoarthritis Outcome Score is a patient assessed outcome score. Questions use a 5 point Likert scale response. KOOS is scored into 5 subscales; Pain, other Symptoms, Activities of Daily Living (ADL) Sport and Recreation Function (Sport/Rec) and knee-related quality of life (QoL). Each subscale ranges from 0 indicating extreme symptoms to 100 indicating no symptoms. Subscale scores will be aggregated and averaged as a primary outcome. The primary analysis repeated measures mixed model will be used to obtain estimates for additional time points as secondary objectives. Changes from baseline of mean subscale scores plotted over time to visualise change.
Change in KOOS -year 7 | baseline (pre-surgery) to year 7 after surgery
  Knee injury and Osteoarthritis Outcome Score is a patient assessed outcome score. Questions use a 5 point Likert scale response. KOOS is scored into 5 subscales; Pain, other Symptoms, Activities of Daily Living (ADL) Sport and Recreation Function (Sport/Rec) and knee-related quality of life (QoL). Each subscale ranges from 0 indicating extreme symptoms to 100 indicating no symptoms. Subscale scores will be aggregated and averaged as a primary outcome. The primary analysis repeated measures mixed model will be used to obtain estimates for additional time points as secondary objectives. Changes from baseline of mean subscale scores plotted over time to visualise change.
Change in KOOS -year 8 | baseline (pre-surgery) to year 8 after surgery
  Knee injury and Osteoarthritis Outcome Score is a patient assessed outcome score. Questions use a 5 point Likert scale response. KOOS is scored into 5 subscales; Pain, other Symptoms, Activities of Daily Living (ADL) Sport and Recreation Function (Sport/Rec) and knee-related quality of life (QoL). Each subscale ranges from 0 indicating extreme symptoms to 100 indicating no symptoms. Subscale scores will be aggregated and averaged as a primary outcome. The primary analysis repeated measures mixed model will be used to obtain estimates for additional time points as secondary objectives. Changes from baseline of mean subscale scores plotted over time to visualise change.
Change in KOOS -year 9 | baseline (pre-surgery) to year 9 after surgery
  Knee injury and Osteoarthritis Outcome Score is a patient assessed outcome score. Questions use a 5 point Likert scale response. KOOS is scored into 5 subscales; Pain, other Symptoms, Activities of Daily Living (ADL) Sport and Recreation Function (Sport/Rec) and knee-related quality of life (QoL). Each subscale ranges from 0 indicating extreme symptoms to 100 indicating no symptoms. Subscale scores will be aggregated and averaged as a primary outcome. The primary analysis repeated measures mixed model will be used to obtain estimates for additional time points as secondary objectives. Changes from baseline of mean subscale scores plotted over time to visualise change.
Change in KOOS - year 10 | baseline (pre-surgery) to year 10 after surgery
  Knee injury and Osteoarthritis Outcome Score is a patient assessed outcome score. Questions use a 5 point Likert scale response. KOOS is scored into 5 subscales; Pain, other Symptoms, Activities of Daily Living (ADL) Sport and Recreation Function (Sport/Rec) and knee-related quality of life (QoL). Each subscale ranges from 0 indicating extreme symptoms to 100 indicating no symptoms. Subscale scores will be aggregated and averaged as a primary outcome. The primary analysis repeated measures mixed model will be used to obtain estimates for additional time points as secondary objectives. Changes from baseline of mean subscale scores plotted over time to visualise change.
Change in Lysholm knee score -week 2 | baseline (pre-surgery) to week 2 after surgery
  Change from baseline as measured by the Lysholm knee score. The Lysholm knee score is a condition-specific outcome measure that contains eight domains: limp, locking, pain, stair-climbing, use of supports, instability, swelling, and squatting. An overall score of 0 to 100 points is calculated, with 95 to 100 points indicating an excellent outcome; 84 to 94 points, a good outcome; 65 to 83 points, a fair outcome; and <65 points, a poor outcome.
Change in Lysholm knee score -week 6 | baseline (pre-surgery) to week 6 after surgery
  Change from baseline as measured by the Lysholm knee score. The Lysholm knee score is a condition-specific outcome measure that contains eight domains: limp, locking, pain, stair-climbing, use of supports, instability, swelling, and squatting. An overall score of 0 to 100 points is calculated, with 95 to 100 points indicating an excellent outcome; 84 to 94 points, a good outcome; 65 to 83 points, a fair outcome; and <65 points, a poor outcome.
Change in Lysholm knee score -month 3 | baseline (pre-surgery) to month 3 after surgery
  Change from baseline as measured by the Lysholm knee score. The Lysholm knee score is a condition-specific outcome measure that contains eight domains: limp, locking, pain, stair-climbing, use of supports, instability, swelling, and squatting. An overall score of 0 to 100 points is calculated, with 95 to 100 points indicating an excellent outcome; 84 to 94 points, a good outcome; 65 to 83 points, a fair outcome; and <65 points, a poor outcome.
Change in Lysholm knee score -month 6 | baseline (pre-surgery) to month 6 after surgery
  Change from baseline as measured by the Lysholm knee score. The Lysholm knee score is a condition-specific outcome measure that contains eight domains: limp, locking, pain, stair-climbing, use of supports, instability, swelling, and squatting. An overall score of 0 to 100 points is calculated, with 95 to 100 points indicating an excellent outcome; 84 to 94 points, a good outcome; 65 to 83 points, a fair outcome; and <65 points, a poor outcome.
Change in Lysholm knee score -year 1 | baseline (pre-surgery) to year 1 after surgery
  Change from baseline as measured by the Lysholm knee score. The Lysholm knee score is a condition-specific outcome measure that contains eight domains: limp, locking, pain, stair-climbing, use of supports, instability, swelling, and squatting. An overall score of 0 to 100 points is calculated, with 95 to 100 points indicating an excellent outcome; 84 to 94 points, a good outcome; 65 to 83 points, a fair outcome; and <65 points, a poor outcome.
Change in Lysholm knee score -year 2 | baseline (pre-surgery) to year 2 after surgery
  Change from baseline as measured by the Lysholm knee score. The Lysholm knee score is a condition-specific outcome measure that contains eight domains: limp, locking, pain, stair-climbing, use of supports, instability, swelling, and squatting. An overall score of 0 to 100 points is calculated, with 95 to 100 points indicating an excellent outcome; 84 to 94 points, a good outcome; 65 to 83 points, a fair outcome; and <65 points, a poor outcome.
Change in Tegner Activity Scale -week 2 | baseline (pre-surgery) to week 2 after surgery
  Change from baseline as measured by the Tegner Activity scale. The Tegner Activity scale contains 11 assessments based on the following domains: competitive sports, recreational sports, work and sick leave. The Tegner activity scale is a one-item score that grades activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer.
Change in Tegner Activity Scale -week 6 | baseline (pre-surgery) to week 6 after surgery
  Change from baseline as measured by the Tegner Activity scale. The Tegner Activity scale contains 11 assessments based on the following domains: competitive sports, recreational sports, work and sick leave. The Tegner activity scale is a one-item score that grades activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer.
Change in Tegner Activity Scale -month 3 | baseline (pre-surgery) to month 3 after surgery
  Change from baseline as measured by the Tegner Activity scale. The Tegner Activity scale contains 11 assessments based on the following domains: competitive sports, recreational sports, work and sick leave. The Tegner activity scale is a one-item score that grades activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer.
Change in Tegner Activity Scale -month 6 | baseline (pre-surgery) to month 6 after surgery
  Change from baseline as measured by the Tegner Activity scale. The Tegner Activity scale contains 11 assessments based on the following domains: competitive sports, recreational sports, work and sick leave. The Tegner activity scale is a one-item score that grades activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer.
Change in Tegner Activity Scale -year 1 | baseline (pre-surgery) to year 1 after surgery
  Change from baseline as measured by the Tegner Activity scale. The Tegner Activity scale contains 11 assessments based on the following domains: competitive sports, recreational sports, work and sick leave. The Tegner activity scale is a one-item score that grades activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer.
Change in Tegner Activity Scale -year 2 | baseline (pre-surgery) to year 2 after surgery
  Change from baseline as measured by the Tegner Activity scale. The Tegner Activity scale contains 11 assessments based on the following domains: competitive sports, recreational sports, work and sick leave. The Tegner activity scale is a one-item score that grades activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer.
Change in Visual Analogue Score (VAS) - week 2 | baseline (pre-surgery) to week 2 after surgery
  Visual Analogue Score - patient assessed pain level where 0 = no pain to 100 = worst imaginable pain. The patient is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity. The measurement from 0 to the line provides a score in the range 0-100mm, with higher scores indicating worse pain. Patients are asked about their current pain or pain intensity in the last 24 hours.
Change in Visual Analogue Score (VAS) - week 6 | baseline (pre-surgery) to week 6 after surgery
  Visual Analogue Score - patient assessed pain level where 0 = no pain to 100 = worst imaginable pain. The patient is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity. The measurement from 0 to the line provides a score in the range 0-100mm, with higher scores indicating worse pain. Patients are asked about their current pain or pain intensity in the last 24 hours.
Change in Visual Analogue Score (VAS) - month 3 | baseline (pre-surgery) to month 3 after surgery
  Visual Analogue Score - patient assessed pain level where 0 = no pain to 100 = worst imaginable pain. The patient is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity. The measurement from 0 to the line provides a score in the range 0-100mm, with higher scores indicating worse pain. Patients are asked about their current pain or pain intensity in the last 24 hours.
Change in Visual Analogue Score (VAS) - month 6 | baseline (pre-surgery) to month 6 after surgery
  Visual Analogue Score - patient assessed pain level where 0 = no pain to 100 = worst imaginable pain. The patient is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity. The measurement from 0 to the line provides a score in the range 0-100mm, with higher scores indicating worse pain. Patients are asked about their current pain or pain intensity in the last 24 hours.
Change in Visual Analogue Score (VAS) - year 1 | baseline (pre-surgery) to year 1 after surgery
  Visual Analogue Score - patient assessed pain level where 0 = no pain to 100 = worst imaginable pain. The patient is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity. The measurement from 0 to the line provides a score in the range 0-100mm, with higher scores indicating worse pain. Patients are asked about their current pain or pain intensity in the last 24 hours.
Change in Visual Analogue Score (VAS) - year 2 | baseline (pre-surgery) to year 2 after surgery
  Visual Analogue Score - patient assessed pain level where 0 = no pain to 100 = worst imaginable pain. The patient is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity. The measurement from 0 to the line provides a score in the range 0-100mm, with higher scores indicating worse pain. Patients are asked about their current pain or pain intensity in the last 24 hours.
Change in EQ-5D-5L -month 6 | baseline (pre-surgery) to month 6 after surgery
  Change from baseline in the EQ-5D-5L score. The EuroQol 5-Dimension 5-Level (EQ-5D-5L) score is a standardised measure of health status developed by the EuroQol Group to provide a simple, generic measure of health for clinical and economic appraisal. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Change in EQ-5D-5L -year 1 | baseline (pre-surgery) to year 1 after surgery
  Change from baseline in the EQ-5D-5L score. The EuroQol 5-Dimension 5-Level (EQ-5D-5L) score is a standardised measure of health status developed by the EuroQol Group to provide a simple, generic measure of health for clinical and economic appraisal. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Change in EQ-5D-5L -year 1 | baseline (pre-surgery) to year 2 after surgery
  Change from baseline in the EQ-5D-5L score. The EuroQol 5-Dimension 5-Level (EQ-5D-5L) score is a standardised measure of health status developed by the EuroQol Group to provide a simple, generic measure of health for clinical and economic appraisal. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Magnetic Resonance Imaging -month 3 | baseline (pre-surgery) to month 3 after surgery
  MRI evaluation of implantation. These scans will allow the assessment of the integrity of the intra-articular structures, the FibroFix™ Cartilage P implant and its integration.
Magnetic Resonance Imaging -month 6 | baseline (pre-surgery) to month 6 after surgery
  MRI evaluation of implantation. These scans will allow the assessment of the integrity of the intra-articular structures, the FibroFix™ Cartilage P implant and its integration.
Magnetic Resonance Imaging -year 1 | baseline (pre-surgery) to year 1 after surgery
  MRI evaluation of implantation. These scans will allow the assessment of the integrity of the intra-articular structures, the FibroFix™ Cartilage P implant and its integration.
Magnetic Resonance Imaging -year 2 | baseline (pre-surgery) to year 2 after surgery
  MRI evaluation of implantation. These scans will allow the assessment of the integrity of the intra-articular structures, the FibroFix™ Cartilage P implant and its integration.
Usability Questionnaire - Surgeons and Theatre nurses | immediately post-surgery
  A usability questionnaire will be completed after performing the surgery to assess their opinion of using the FibroFix Cartilage P implant and Drill set by surgeons and theatre nurses.
  The data collected may be from open questions or using Likert scales to determine the strength of opinion. Analysis of the data collected during the formative evaluations and summative testing will be presented in the form of descriptive summaries, diagrammatic form (e.g., bar charts or histograms), and simple computation calculations such as means, standard deviations where possible, ranges of results, or percentages (e.g., percentage of people that thought…).
Usability Questionnaire - Processing staff | after processing of instruments
  A usability questionnaire will be completed by the processing staff after processing (cleaning and sterilizing) the Drill set (instrumentation used to prepare the implant site during surgery) to assess their opinion of the ease of cleaning and sterilizing the instruments.
  The data collected may be from open questions or using Likert scales to determine the strength of opinion. Analysis of the data collected during the formative evaluations and summative testing will be presented in the form of descriptive summaries, diagrammatic form (e.g., bar charts or histograms), and simple computation calculations such as means, standard deviations where possible, ranges of results, or percentages (e.g., percentage of people that thought…).
Usability Questionnaire - Patients | pre-discharge from hospital
  A usability questionnaire will be completed by the Patients after being given the implant card and related patient leaflet after surgery and before discharge to assess their opinion of the ease of understanding of the material given to them.
  The data collected may be from open questions or using Likert scales to determine the strength of opinion. Analysis of the data collected during the formative evaluations and summative testing will be presented in the form of descriptive summaries, diagrammatic form (e.g., bar charts or histograms), and simple computation calculations such as means, standard deviations where possible, ranges of results, or percentages (e.g., percentage of people that thought…).
Safety endpoint - month 3 | up to month 3 after surgery
  Cumulative incidence of device-related Adverse Events
Safety endpoint - month 6 | up to month 6 after surgery
  Cumulative incidence of device related Adverse Events
Safety endpoint -year 2 | up to year 2 after surgery
  Cumulative incidence of device related Adverse Events
Safety endpoint -year 3 | up to year 3 after surgery
  Cumulative incidence of device related Adverse Events
Safety endpoint -year 4 | up to year 4 after surgery
  Cumulative incidence of device related Adverse Events
Safety endpoint -year 5 | up to year 5 after surgery
  Cumulative incidence of device related Adverse Events
Safety endpoint -year 6 | up to year 6 after surgery
  Cumulative incidence of device related Adverse Events
Safety endpoint -year 7 | up to year 7 after surgery
  Cumulative incidence of device related Adverse Events
Safety endpoint -year 8 | up to year 8 after surgery
  Cumulative incidence of device related Adverse Events
Safety endpoint -year 9 | up to year 9 after surgery
  Cumulative incidence of device related Adverse Events
Safety endpoint -year 10 | up to year 10 after surgery
  Cumulative incidence of device related Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Michael Whitehouse, Principal Investigator — North Bristol NHS HospitalsTrust
Locations (2):
- Menta Egészségközpont, Budapest, Hungary
- North Bristol NHS Trust, Bristol, United Kingdom